CLINICAL TRIAL: NCT03418272
Title: Oral and Tracheal Cultures in Pediatric ICU Patients Compared to Healthy Children
Brief Title: Cultures in PICU Patients Compared to Healthy Children
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn until time and staff allow its completion.
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Christopher Heard, Clinical Professor of Anesthesiology, State University of New York at Buffalo
Other Study IDs: STUDY00001954
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Ventilator Associated Pneumonia; Pneumonia, Bacterial
Keywords: ICU; OR; Pneumonia; PICU; Pediatric; PCR
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia, Bacterial; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ventilated Pediatric Intensive Care Unit patient Group: This will be a prospective descriptive case series where tracheal cultures and PCR results will be analyzed at initial intubation and again several days into the ICU stay.
  Interventions: Diagnostic Test: Culture/PCR Analysis
- Intubated OR patient Control Group: For the healthy operating room children, also a case series where a single set of studies will be obtained. tracheal cultures and PCR results will be analyzed after intubation These two groups will be compared, non-randomized.
  Interventions: Diagnostic Test: Culture/PCR Analysis

INTERVENTIONS:
Diagnostic Test: Culture/PCR Analysis — Microbes to be selectively cultured and PCR analysis to be conducted. Bacteria obtained in samples will be dispersed in non-selective Mueller Hinton Broth (Sigma-Aldrich), divided into two separate cultures and grown overnight at 37°C in aerobic condition and in 5% CO2 to assure survival of both aerobic and facultative anaerobic species.
  * Staphylococcus aureus (MSSA, MRSA)
  * Pseudomonas aeruginosa
  * Haemophilus influenza
  * Streptococcus pneumonia
  * Streptococcus Pyogenes Group B streptococci,
  * Klebsiella pneumonia
  * Moraxella catarrhalis

SUMMARY:
This study is being done to determine if the bacteria found in your mouth (oral flora bacteria) in children admitted to the intensive care unit who need to be on a breathing machine is different from the oral flora in healthy children undergoing anesthesia for their dental caries. Children in the intensive care unit with a breathing tube are at a higher risk for getting a lung infection due to the bacteria in the mouth slipping into their lungs past the breathing tube over several days. This means that bacteria are found in the child's lung when this is normally not the case. If the bacteria in the mouth have changed from normal then they may get a pneumonia.

DETAILED DESCRIPTION:
The oral cavity has natural flora of microbiology that may be associated with the development of dental decay. Another possible problem arising from this flora is the migration of the bacteria into the trachea causing pulmonary infections such as trachietis or pneumonia. The risk of developing a pulmonary infection appears to be increased in patients who have been intubated for a period of time (days) such as those patients ventilated in the intensive care unit (ICU). It has also been shown that in patients in the ICU the nature of the oral flora changes over time to include bacteria that are more commonly associated with the nosocomial pneumonia, ventilator associated pneumonia. We have previous demonstrated in a small pilot study (CYIRB2779) that the changes in the oral flora in children intubated in the ICU was similar to those bacteria grown from tracheal cultures ordered by the intensivist. Patients intubated in the ICU maybe at risk of decreased salivary flow, sedated and unable to clear secretions and are reliant on the bedside nurse to maintain adequate oral hygiene. Most ICU's have guidelines and policies to ensure that oral hygiene is appropriately cared for. They are also at risk for changes in the oral flora due to concomitant broad-spectrum antibiotic use that is common in the initial 48 hours after admission with respiratory failure.

The second are of interest is to determine whether children who are very sick and require intubation and ventilation support have different bugs growing in their mouth that may predispose them to future infection whilst in the ICU.

ELIGIBILITY:
Inclusion Criteria:

ICU Group:

* Intubated within 12 hours
* ASA 1 or 2 (ASA - AMERICAN SOCIETY ANESTEHESIOLOGY PREOPOERATIVE STATUS)
* Age 2 to 8

OR Group:

* ASA 1 or 2
* Elective dental surgery requiring intubation
* Age 2 to 8

Exclusion Criteria:

ICU Group:

* Trauma patients
* Postoperative patients
* Children under 2 or over 8

OR Group:

* Received antibiotics within the last week
* Received prednisone within the last 2 weeks
* Viral respiratory infective process within the last 2 weeks

Ages: 2 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: ICU Group:
  * Intubated within 12 hours
  * ASA 1 or 2 (ASA - AMERICAN SOCIETY ANESTEHESIOLOGY PREOPOERATIVE STATUS)
  * Age 2 to 8
  OR Group:
  * ASA 1 or 2
  * Elective dental surgery requiring intubation
  * Age 2 to 8
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of bacteria in sample | By January 2019
  PCR analysis
Presence of bacteria in sample | By January 2019
  Culture analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Heard, MBChB, FRCA, Principal Investigator — Jacobs School of Medicine

IPD SHARING:
Plan to Share IPD: No